CLINICAL TRIAL: NCT00284492
Title: Effectiveness of Acupuncture-care for Treatment of Hot Flushes Among Postmenopausal Women
Brief Title: Acupuncture for Hot Flushes in Menopause
Acronym: ACUFLASH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of North Norway (Other)
Collaborators: The Research Council of Norway (Other); University of Tromso (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P REK NORD 102/2005
Record Dates: First submitted 2006-01-30; First posted 2006-01-31 (Estimated); Last update posted 2012-05-14 (Estimated); Status verified 2012-05

CONDITIONS: Menopause; Hot Flashes
Keywords: Women; Acupuncture; Menopause; Hot flashes; Health related quality of life
MeSH Terms: conditions — Hot Flashes | interventions — Self Care

ARMS (2):
- Lifestyle advice (Active Comparator)
  Interventions: Behavioral: Self Care
- Lifestyle advice and acupuncture therapy (Experimental)
  Interventions: Procedure: Traditional chinese medicine type acupuncture

INTERVENTIONS:
Procedure: Traditional chinese medicine type acupuncture — 10 acupuncture sessions
  Arms: Lifestyle advice and acupuncture therapy
Behavioral: Self Care — Lifestyle advice on diet, physical activity
  Arms: Lifestyle advice

SUMMARY:
In a pragmatic study investigate whether Traditional Chinese Medicine acupuncture-care decreases the frequency of hot flushes and increases health related quality of life among postmenopausal women. The intervention group will receive 10 sessions of acupuncture, the control group will engage in self care only. The study period lasts for 12 weeks.

DETAILED DESCRIPTION:
The study objective is to determine whether Traditional Chinese Medicine (TCM) acupuncture-care together with self-care is more effective than self-care alone, to relieve climacteric complaints among women who seek alternatives to hormonal replacement therapy (HRT). Study design is a pragmatic randomised controlled trial with two parallel arms. Study participants are postmenopausal women who document a mean value of 7 flushes/24 hours and who are not using HRT or other prescribed medication that may influence climacteric complaints. The treatment group will receive 10 sessions of TCM acupuncture-care and self-care; the control group will engage in self-care only.

The duration of intervention period is 12 weeks with evaluations at baseline, 4, 8, 12 weeks, and follow up at 6 and 12 months after baseline. Primary endpoint is change in daily hot flush frequency in the two groups from baseline to 12 weeks; secondary endpoint is health related quality of life. N in each treatment group: 143 (286 altogether).

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women (at least one year past the last menstrual period) who are willing to receive acupuncture and who during two weeks of self-completed diaries10 document a mean value of 7 flushes/24 hours or more (or 50 flushes or more over a period of seven consecutive days), will be randomized after a baseline evaluation.
* Current users prescribed medications that influence hot flush rate (e. g. HRT, SSRI's) can be included after a washout period. The washout-periods are eight weeks for SSRI's and systemic (including transdermal) HRT and four weeks for local estradiol preparations

Exclusion Criteria:

* Surgical menopause
* History of cancer within the past five years
* Use of anticoagulant drugs
* Heart valve disease
* Poorly controlled hypertension
* Hypothyroidism
* Hyperthyroidism or diabetes mellitus
* Organ transplant
* Mental disease
* Overt drug or alcohol dependency
* Inability to complete study forms

Ages: 40 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 286 (Actual)
Dates: Start 2006-02; Primary Completion 2007-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Frequency of hot flushes | 12 weeks

SECONDARY OUTCOMES:
Health related quality of life (Women's Health Questionnaire) | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sameline Grimsgaard, MD, MPH, PhD, Principal Investigator — University Hospital of North Norway. No-9038 Tromsø, Norway
Locations (1):
- Clinical Research Center, University Hospital of North Norway, Tromsø, Norway